CLINICAL TRIAL: NCT05250128
Title: Characterization and Significance of Circulating Microvesicles in Pulmonary Hypertension Due to Chronic Obstructive Pulmonary Disease
Brief Title: The Significance of Circulating Microvesicles in Pulmonary Hypertension Due to Chronic Obstructive Pulmonary Disease
Acronym: MICROBOPH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8073
Record Dates: First submitted 2022-02-04; First posted 2022-02-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-02

CONDITIONS: Pulmonary Hypertension Due to Chronic; Obstructive Pulmonary Disease; Circulating Microvesicles; Circulating Markers of Endothelium Damage
MeSH Terms: conditions — Lung Diseases, Obstructive | interventions — Catheterization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — During right-heart catheterization, blood samples are collected from the occluded pulmonary artery and the jugular vein.
  Platelet-poor plasma (PPP) samples are obtained by double centrifugation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Catheterization — Right heart catheterization, using the Swan-Ganz standard technique, to measure mean pulmonary arterial pressure, pulmonary capillary wedge pressure, cardiac output and pulmonary vascular resistance

SUMMARY:
Mild to moderate pulmonary hypertension is a common complication of chronic obstructive pulmonary disease (COPD); such a complication is associated with increased risks of exacerbation and decreased survival. A small proportion of COPD patients may present with severe pulmonary hypertension, defined by a mean pulmonary artery pressure more than 35 mmHg (or more than 20 mmHg with a low cardiac index < 2 l/min/m2) with pulmonary vascular resistance more than 3 Wood units, measured by right heart catheterization (RHC). In these patients, pulmonary microvessels remodeling is the main cause of increase in pulmonary arterial pressure and is thought to result from the combined effects of hypoxia, inflammation, and loss of capillaries but the mechanisms are complex.

For these patients, no drugs have been approved for treatment and lung transplantation must be considered for the more severe patients who are eligible. A better characterization of these patients is needed.

We hypothesize that microvesicles generation and endothelial damage could be related to the severity of pulmonary hypertension due to COPD, assessed by pulmonary hemodynamic parameters. Circulating biomarkers of vascular damage and cell activation will be measured in blood samples from 80 COPD patients who have hemodynamic assessment by RHC. To go further, the origin of the particles will be characterized.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18
* COPD: obstructive ventilatory insufficient on spirometry and history of smoking
* patients who will perform right heart catheterization
* Signature of written informed consent

Exclusion criteria:

* LVEF < 45% (echocardiography)
* Post-capillary pulmonary hypertension (pulmonary capillary wedge pressure > 15 mmHg)
* Chronic Thromboembolic hypertension
* Pulmonary embolism < 6 months
* Acute coronary syndrome < 3 months
* Significant cardiac valvulopathy (echocardiography)
* Portal hypertension
* Connective tissue disease
* chronic renal insufficient (clearance < 40 ml/min)
* Glycated hemoglobin > 7% (if diabetes)
* Non controlled arterial hypertension
* Positive beta-HCG
* Respiratory exacerbation during the inclusive period
* Patients under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic obstructive pulmonary disease, addressed to the competence center PulmoTension of the Strasbourg University hospital, France:
  * who are considered for lung transplantation;
  * with severe hypoxemia;
  * with suspicion of pulmonary hypertension (on echocardiography) And who perform right heart catheterization.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Study the rate of circulating endothelial microparticles (EPPs) according to the severity of pulmonary hypertension associated with COPD. | - During the first hemodynamic assessment by RHC; - At 3 to 6 months, if hemodynamic control is required (RHC)
  Circulating biomarkers of vascular damage and cell activation will be measured in blood samples from COPD patients who have hemodynamic assessment by RHC. Samples will be withdrawn from occluded pulmonary artery and jugular vein during the exam.

SECONDARY OUTCOMES:
Characterization of circulating microvesicles in pulmonary hypertension due to chronic obstructive pulmonary disease | - During the first hemodynamic assessment by RHC; - At 3 to 6 months, if an hemodynamic control is required (RHC)
  Circulating markers of endothelium damage with circulating microvesicles will be dosed.
Characterization of circulating microvesicles in pulmonary hypertension due to chronic obstructive pulmonary disease | - During the first hemodynamic assessment by RHC; - At 3 to 6 months, if an hemodynamic control is required (RHC)
  Proinflammatory markers with circulating microvesicles will be dosed.
Characterization of circulating microvesicles in pulmonary hypertension due to chronic obstructive pulmonary disease | - During the first hemodynamic assessment by RHC; - At 3 to 6 months, if an hemodynamic control is required (RHC)
  Cell stimulation estimated with circulating microvesicles will be dosed.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne RIOU, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaire de Strasbourg - Service Pneumologie - centre de compétence de l'hypertension artérielle pulmonaire - France, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided